CLINICAL TRIAL: NCT04948073
Title: The Effects of Dynamic Neuromuscular Stabilization Approach on Functional Movement Patterns, Balance, Quality of Life, and Exercise Capacity in Older Patients With Chronic Nonspecific Low Back Pain
Brief Title: The Effects of Dynamic Neuromuscular Stabilization Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, Caner Karartı, Hacettepe University, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021500
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain; Rehabilitation; Treatment
Keywords: low back pain; rehabilitation; stabilization; exercises; balance
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Outcomes Assessor
Masking Description: the blinded assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will follow a DNS exercise protocol based on previous procedure for a whole period of 6 weeks (three 50-min sessions per week) in addition the conventional treatment. DNS group's protocol will involve 5 min warm-up, 40 min DNS movements (4 different parts, each part lasts for 10 min) accompanied with breathing exercises, and 5 min cool-down. DNS exercises will include diaphragmatic breathing, Baby Rock, Rolling, Side Lying, Oblique Sit, Tripod, Kneeling, Squat, Prone, and Czech Get Up (CGU). Week one specifically will involve training and practicing basic DNS exercises. The complexity of the exercises will increase gradually by adding a new task to an already practiced task every week. An increase in the complexity of a task will help the performer to automate performance. We will use the dual-task paradigm to examine if the task is automated or not (e.g. no new task should disturb the diaphragmatic breathing).
  Interventions: Other: Dynamic neuromuscular stabilization approach
- Control Group (Active Comparator): Patients from both groups will receive a conventional 6-week treatment programme (18 treatment sessions, three a week, for 30-40min duration). All patients will also continue their usual activities and receive advices related to the daily living activites in the form of a leaflet. Participants will be asked to refrain from seeking any other types of rehabilitation treatments during the trial. The conventional physical therapy program for both groups includes: TENS therapy for the low back (15 min 3 days/week), with a frequency of 100 Hz and fixed pulse; ultrasound for 5 minutes, 1 Hz, continuous mode of application 1.5 w/cm2. The exercise programs will consist strengthening, stretching exercises for the abdominal, back, pelvic, and lower limb muscles.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Dynamic neuromuscular stabilization approach — The experimental group will follow a DNS exercise protocol based on previous procedure for a whole period of 6 weeks (three 50-min sessions per week) in addition the conventional treatment.
  Arms: Experimental Group
Other: Conventional treatment — Patients from both groups will receive a conventional 6-week treatment programme (18 treatment sessions, three a week, for 30-40min duration).
  Arms: Control Group

SUMMARY:
When the positive effects of the recently popular "Dynamic Neuromuscular Stabilization (DNS)" approach are examined, it suggests that it may be a possible treatment option in geriatric individuals with chronic nonspecific low back pain (CSNLP). Based on the principles of developmental kinesiology, the DNS approach takes advantage of infants' motor development curves in the treatment of motor disorders. The main focus is on regulating intra-abdominal pressure and the integrated spinal stabilizing system (ISSS) through specific functional exercises based on the positions exhibited by a healthy infant. According to the DNS, every developmental position is an exercise position, but every exercise must follow basic principles. These principles are restoration of correct respiratory pattern and intra-abdominal pressure, respectively; ensuring correct support during dynamic activities of the extremities and ensuring biomechanical alignment during movement. Considering the principles of exercise, there appears to be a potential mechanism of action for anomalies in geriatric individuals with CNSLBP. Therefore, in our study, we aimed to examine the effect of DNS approach on functional movement patterns, balance, quality of life and exercise capacity in geriatric individuals with CNSLBP. It is the first randomized controlled study in the literature, and our hypothesis is that the DNS approach may be an effective therapeutic approach on these parameters.

DETAILED DESCRIPTION:
It has been reported that during isometric upper and lower extremity flexion exercises in individuals with chronic nonspecific low back pain (CSNLP), the mobility of the diaphragm decreases, especially in the anterior-middle portions. The regulation of intra-abdominal pressure is impaired due to insufficient mobility of the diaphragm and causes compressive forces on the vertebrae due to the compensatory activity of the superficial spinal extensors. Muscle imbalance between the upper and lower quadrants also results in an abnormal position of the chest or rib cage, negatively affecting lung function and exercise capacity. When the positive effects of the recently popular "Dynamic Neuromuscular Stabilization (DNS)" approach are examined, it suggests that it may be a possible treatment option in geriatric individuals with CSNLP. Based on the principles of developmental kinesiology, the DNS approach takes advantage of infants' motor development curves in the treatment of motor disorders. The main focus is on regulating intra-abdominal pressure and the integrated spinal stabilizing system through specific functional exercises based on the positions exhibited by a healthy infant. According to the DNS, every developmental position is an exercise position, but every exercise must follow basic principles. These principles are restoration of correct respiratory pattern and intra-abdominal pressure, respectively; ensuring correct support during dynamic activities of the extremities and ensuring biomechanical alignment during movement. Considering the principles of exercise, there appears to be a potential mechanism of action for anomalies in geriatric individuals with CNSLBP. Therefore, in our study, we aimed to examine the effect of DNS approach on functional movement patterns, balance, quality of life and exercise capacity in geriatric individuals with CNSLBP. It is the first randomized controlled study in the literature, and our hypothesis is that the DNS approach may be an effective therapeutic approach on these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being an older patient seeking care for CNSLBP (with a duration of at least 3 months) without leg pain.
* To have a pain intensity of at least 3 points (measured on a 0-10 point Visual Analog Scale (VAS);
* The ability to comprehend and follow verbal instructions,
* To be over 65 years of age,
* To volunteer to participate in the study

Exclusion Criteria:

* history of spinal surgery
* severe spinal pathologies (e.g. ankylosing spondylitis, lumbar spinal stenosis, spina bifida, spinal tumors, osteoporosis, and cauda equina syndrome)
* medical contraindications to active exercise;
* concomitant somatic or psychiatric disorder [Mini-Mental State Examination score ≤24]
* neurological deficits (e.g. brain tumor and nerve palsies); specific causes of LBP (e.g. facet joint problem, disc herniation, sacroiliac joint dysfunction)
* nerve root compression
* spinal deformities
* autoimmune diseases (e.g. rheumatoid arthritis and systemic lupus erythematosus)
* cancer

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screening (FMS) [Functional Movement Patterns) | 6 weeks
  FMS will be used to evaluate the quality of 7 functional movement patterns with the goal of identifying movement limitations and asymmetries. The FMS consists of 7 individual test items including the deep squat, in-line lunge, hurdle step, shoulder flexibility, push-up, straight leg raise, and rotary trunk stability assessment. Each of these 7 test items is graded on a scale of 0-3; thus, the lowest and highest possible overall FMS scores are 0 and 21, respectively.
6-Minute Walk Test (6MWT) [Exercise Capacity] | 6 weeks
  6MWT is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes.It provides information regarding functional capacity, response to therapy and prognosis across a broad range of chronic cardiopulmonary conditions. Main strengths of the 6MWT stem from its simplicity in concept and performance, low cost, ease of standardization, and acceptance by test subjects, including those who are deconditioned, elderly, or frail.

SECONDARY OUTCOMES:
Timed-up and go Test (TUG) [Balance] | 6 weeks
  TUG is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally require. The TUG is used frequently in the elderly population, as it is easy to administer and can generally be completed by most older adults.
WHOQOL-OLD module [Quality of life] | 6 weeks
  It consists of 24 items assigned to 6 dimensions, the responses to which are determined by the five-level Likert scale. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolar P, Sulc J, Kyncl M, Sanda J, Cakrt O, Andel R, Kumagai K, Kobesova A. Postural function of the diaphragm in persons with and without chronic low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):352-62. doi: 10.2519/jospt.2012.3830. Epub 2011 Dec 21. PMID 22236541
- [Background] Scott S, Fuld JP, Carter R, McEntegart M, MacFarlane NG. Diaphragm ultrasonography as an alternative to whole-body plethysmography in pulmonary function testing. J Ultrasound Med. 2006 Feb;25(2):225-32. doi: 10.7863/jum.2006.25.2.225. PMID 16439786
- [Background] Kolar P, Neuwirth J, Sanda J, Suchanek V, Svata Z, Volejnik J, Pivec M. Analysis of diaphragm movement during tidal breathing and during its activation while breath holding using MRI synchronized with spirometry. Physiol Res. 2009;58(3):383-392. doi: 10.33549/physiolres.931376. Epub 2008 Jul 18. PMID 18637703
- [Background] Kolar P, Sulc J, Kyncl M, Sanda J, Neuwirth J, Bokarius AV, Kriz J, Kobesova A. Stabilizing function of the diaphragm: dynamic MRI and synchronized spirometric assessment. J Appl Physiol (1985). 2010 Oct;109(4):1064-71. doi: 10.1152/japplphysiol.01216.2009. Epub 2010 Aug 12. PMID 20705944
- [Background] Mahdieh L, Zolaktaf V, Karimi MT. Effects of dynamic neuromuscular stabilization (DNS) training on functional movements. Hum Mov Sci. 2020 Apr;70:102568. doi: 10.1016/j.humov.2019.102568. Epub 2020 Jan 13. PMID 31950895
- [Background] Son MS, Jung DH, You JSH, Yi CH, Jeon HS, Cha YJ. Effects of dynamic neuromuscular stabilization on diaphragm movement, postural control, balance and gait performance in cerebral palsy. NeuroRehabilitation. 2017;41(4):739-746. doi: 10.3233/NRE-172155. PMID 29254112
- [Background] Yoon HS, Cha YJ, You JSH. Effects of dynamic core-postural chain stabilization on diaphragm movement, abdominal muscle thickness, and postural control in patients with subacute stroke: A randomized control trial. NeuroRehabilitation. 2020;46(3):381-389. doi: 10.3233/NRE-192983. PMID 32250328
- [Background] Inani SB, Selkar SP. Effect of core stabilization exercises versus conventional exercises on pain and functional status in patients with non-specific low back pain: a randomized clinical trial. J Back Musculoskelet Rehabil. 2013;26(1):37-43. doi: 10.3233/BMR-2012-0348. PMID 23411647